CLINICAL TRIAL: NCT01250327
Title: Medico-economic Evaluation of a Non-chirurgical Pulmonary Valve Replacement for the Treatment of Lesions of the Ventricular Outflow Tract.
Brief Title: Medico-economic Evaluation of a Non-chirurgical Pulmonary Valve Replacement (REVALV)
Acronym: REVALV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P080205
Record Dates: First submitted 2010-11-27; First posted 2010-11-30 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Dysfunction of the Prosthetic Conduct; Lesions of the Right Ventricular Outflow Tract
Keywords: right ventricular outflow tract; endovascular valve insertion; economic evaluation; valved stent
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Melody (Experimental): insertion of a pulmonic valved stent
  Interventions: Device: Melody
- Bare stent (Active Comparator): insertion of a bare metal stent
  Interventions: Device: bare stent
- Surgery (Active Comparator): conventional surgery methode.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Device: Melody — insertion of a pulmonic valved stent
  Other Names: insertion of a pulmonic valved stent
  Arms: Melody
Device: bare stent — insertion of a bare metal stent
  Other Names: insertion of a bare metal stent
  Arms: Bare stent
Procedure: Surgery — conventional surgery methode
  Other Names: conventional surgery methode
  Arms: Surgery

SUMMARY:
This prospective interventional study is designed to evaluate the cost/advantage ratio in the treatment of lesions of the right ventricular outflow tract using transcatheter pulmonary valved stent (Melody).

DETAILED DESCRIPTION:
Rational : transcatheter valve insertion is a new technique enlarging the armamentarium of the treatment of RVOT obstruction and insufficiency. It real place as compared to bare stent implantation and surgery of the RVOT remains unknown.

Main objective : evaluate the cost of the procedure as compared with conventional technique.

Design : multicenter intervention prospective study. Population : 180 patients in three arms (3*60).

End point criteria :

* Primary : cost
* Secondary : rate of reoperation

ELIGIBILITY:
Inclusion Criteria:

for the study:

* Lesions of the right ventricular outflow tract in need of surgery for stenosis or regurgitation

for the Melody arm:

* A 5 to 70 years old patient
* Weight >= 30kg
* RVOT <= to 22mm
* Patient with a dysfunction circumferential prosthetic conduct of diameter >= to 16mm.

Exclusion Criteria:

* Vein anatomy incompatibility with a 22Fr delivery health
* Left heart implantation
* RVOT incompatible with a anchoring of the stent (lik in patient operated of a tetralogy of fallot)
* Coronary anomaly with a coronary artery naer the RVOT
* Sever obstruction of the RVOT incompatible with balloon expansion
* Central vein obstruction
* Ongoing infection
* Active endocarditis
* Allergy for heparin or aspirin
* Pregnancy

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2009-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Cost induced by the transcatheter pulmonary valve insertion as compared to conventional surgical and insertion of a bare metal stent 24 months after insertion. | 24 months after intervention

SECONDARY OUTCOMES:
Quality of life | 24 months after intervention
procedure success rate | 24 months after intervention
Does the patient need to be operated again? | 24 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Boudjemline Younes, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Necker Enfants Malades, Paris, France

REFERENCES:
- [Derived] Fraisse A, Aldebert P, Malekzadeh-Milani S, Thambo JB, Piechaud JF, Aucoururier P, Chatelier G, Bonnet D, Iserin L, Bonello B, Assaidi A, Kammache I, Boudjemline Y. Melody (R) transcatheter pulmonary valve implantation: results from a French registry. Arch Cardiovasc Dis. 2014 Nov;107(11):607-14. doi: 10.1016/j.acvd.2014.10.001. Epub 2014 Nov 6. PMID 25453718